CLINICAL TRIAL: NCT05154370
Title: China National Registry of Neuro-Inflammatory Diseases: a Prospective Cohort Study
Brief Title: China National Registry of Neuro-Inflammatory Diseases
Acronym: CNRID
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2021-150-01
Record Dates: First submitted 2021-11-08; First posted 2021-12-13 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis; NMO Spectrum Disorder; Clinically Isolated Syndrome; CNS Demyelinating Autoimmune Diseases; Acute Disseminated Encephalomyelitis; Primay Angiitis of the Central Nervous System; Autoimmune Glial Fibrillary Acidic Protein Astrocytopathy
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica; Demyelinating Autoimmune Diseases, CNS; Encephalomyelitis, Acute Disseminated | interventions — Immunoglobulins; Antirheumatic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and cerebral spinal fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

GROUPS / COHORTS (4):
- MS/CIS: Diagnosis of MS and CIS based on the 2017 McDonald MS diagnostic criteria.
  Interventions: Drug: Intravenous steroid
- ADEM: Diagnosis of ADEM based on the 2012 IPMSSG diagnostic criteria for ADEM
  Interventions: Drug: Intravenous steroid
- MOGAD: Diagnosis of MOGAD based on the 2020 Chinese Expert Consensus.
  Interventions: Drug: Intravenous steroid
- NMOSD: diagnosis of NMOSD according to 2015 International Panel for Neuromyelitis Optica Diagnosis criteria.
  Interventions: Drug: Intravenous steroid

INTERVENTIONS:
Drug: Intravenous steroid — This study does not limit treatment methods. Patients commonly use high-dose intravenous steroid therapy (HD-S) during acute stage. Immunomodulatory therapies are necessary for the remission stage. All drugs are used in accordance with relevant guidelines.
  Other Names: Immunoglobulin; Immunosuppressive Drugs; Disease-Modifying Drugs

SUMMARY:
Central nervous system (CNS) idiopathic inflammatory demyelinating diseases (IDD) are mainly diseases caused by autoimmune factors that result in CNS demyelination damage and loss. It tends to accumulate in the brain, spinal cord and optic nerves. Multiple sclerosis (MS), clinically isolated syndrome (CIS), neuromyelitis optica spectrum disorder (NMOSD), myelin oligodendrocyte glycoprotein antibody-associated disease (MOGAD) and acute disseminated encephalomyelitis (ADEM) are all common IDDs of the CNS. Besides, primary angiitis of the central nervous system (PACNS), autoimmune glial fibrillary acidic protein astrocytopathy (GFAP-A), etc. may also be included because they are important differential diagnoses. This study will establish a large prospective cohort study database of Chinese IDD, which will record detailed electronic information on IDD patients, including demographic and socioeconomic data, medical history, clinical information, medication, and relevant examination results. The long-term observational study will be used to understand the natural history of disease, disability progression rates, imaging and biological indicators, long-term treatment approaches and prognosis of Chinese patients with IDD, to find predictive markers for IDD progression and prognosis, and to identify factors that influence the treatment and prognosis of patients with IDD.

DETAILED DESCRIPTION:
Large prospective cohort studies allow long-term observation and analysis of the clinical status and disease activity of IDD patient population, and are the best way to understand IDD's natural course, clinical outcome, and drug efficacy in specific populations. Globally, several large prospective follow-up cohort studies have been conducted, providing important information on the disease characteristics of IDD patients. However, there is no large nationwide registry study of CNS IDD in China, and therefore there is a relative lack of data on the natural course of disease and drug efficacy in the Chinese IDD patient population, as well as a lack of standardized follow-up management of Chinese IDD patients. This study will establish a large prospective cohort study database of Chinese IDD, which will record detailed electronic information on IDD patients. We aim to establish a national (multicenter) disease registry for central nervous system idiopathic inflammatory demyelinating diseases in China, and to establish a unified standardized follow-up management process and treatment guidelines for patients with IDD in China; To provide real world data on the disease status of Chinese IDD patients; To understand the disease progression characteristics of IDD in China; To search for biological and imaging markers that predict the relapse, progression, and prognosis of IDD; to investigate the efficacy, safety, compliance and switch of different disease-modifying drugs (DMDs) in the long-term treatment of Chinese patients with IDD.

The study is a prospective observational (non-interventional) national multicenter cohort study to collect clinical data from IDD patients who have signed informed consent, to routinely and regularly follow up IDD patients on multiple clinical indicators, and to assess clinical outcomes. All information is to be completed prospectively from the time point the patient visited the hospital (except for Basic patient information and information about previous disease that are required at enrollment follow-up).Once the project started, the study sites are not allowed to discontinue the study on their own until the end of study is announced. In addition, to ensure the continuity of the data, each site needs to appoint designated clinical data collectors to collect data from qualified inpatient clinical cases consecutively, so as to ensure the consecutive registration of each inpatient case who meets the inclusion and exclusion criteria.

As the purpose of this study is to establish a national multicenter disease registry to provide disease-related information on patients with IDD in China, and the primary and secondary endpoints of the study being descriptive endpoints, therefore no formal calculation of sample size is needed. 10000 IDD patients are planned to be recruited.

ELIGIBILITY:
Inclusion Criteria:

* 1. No requirement for age and sex
* 2. Need to meet the diagnosis of at least one IDD (clinically isolated syndrome (CIS)/multiple sclerosis (MS)/neuromyelitis optica spectrum disorder (NMOSD)/MOG antibody-associated disease (MOGAD)/acute disseminated encephalomyelitis (ADEM).
* 3. Signed informed consent form.

Exclusion Criteria:

* Those with severe mental disease unable to cooperate with the examination and/or follow-up.
* Any patient (or the patient's legal representative) who is unable or refuses to sign informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 10000 IDD patients are planned to be recruited from many sites throughout the country.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Annual relapse rate (ARR) between baseline and follow-up in patients with IDD | baseline up to 5 years
  a new neurological worsening lasting for at least 24 hours and occurring more than 30 days after the previous attack.
Change in EDSS scores of patients with IDD between baseline and follow-up over time | baseline, Month 6, Month12, Month18, Month24, Month30, Month36, Month42, Month48, Month54, Month60
  The Expanded Disability Status Scale (EDSS) is a rating system that is frequently used for classifying and standardizing the severity and progression. EDSS ranges from 0 to 10. The higher the score, the worse the clinical symptoms.

SECONDARY OUTCOMES:
The brain structural change over time between the baseline MRI and the follow-up MRIs | baseline, year1, year2, year3, year4, year5.
  To describe changes of lesions, grey matter and white matter in patients with neuroinflammatory and demyelination disease measured by Brain Magnetic Resonance Imaging (MRI). The MRI sequence includes T2W_TRA、DWI、3DT1W_TFE_SAG、fMRI_EPI_TRA、mb2DKI_iso48_b1k2k_TRA、3DFLAIR_TSE_SAG、3DpCASL_GRASE_TRA、3DDIR_SAG、3DT2W_TSE、SWI_QSM_TRA. The secondary endpoint is the change over time between the baseline MRI and the follow-up MRIs, of the lesions and brain volumes.
The spinal cord change over time between the baseline MRI and the follow-up MRIs. | baseline, year1, year2, year3, year4, year5.
  To describe changes of lesions and integrity of fiber bundle in spinal cord in neuroinflammatory and demyelination disease patients measured by MRI. The primary endpoint is the change over time between the baseline MRI and the follow-up MRIs, of structural change in spinal cord.
Change of the central vein sign at 7T MRI. | baseline, year1, year2, year3, year4, year5.
  The central vein sign has been proposed as a specific imaging biomarker for distinguishing between multiple sclerosis (MS) and not MS.
Change of rim of iron at 7T MRI. | baseline, year1, year2, year3, year4, year5.
  multiple sclerosis white matter lesions surrounded by a rim of iron containing microglia, termed iron rim lesions, signify patients with more severe disease course and a propensity to develop progressive multiple sclerosis.
Change in High-contrast Letter Acuity (HCLA) over time at baseline and during follow-up in patients with IDD | baseline, year1, year2, year3, year4, year5.
  Adjusted mean change in HCLA every year from baseline as determined by 100% high contrast Sloan letter charts, adjusted for the baseline HCLA value.
Change in Low-contrast Letter Acuity (LCLA) over time at baseline and during follow-up in patients with IDD | baseline, year1, year2, year3, year4, year5.
  Adjusted mean change in LCLA at baseline and every year as determined by 2.5% low contrast Sloan letter charts，adjusted for the baseline LCLA value.
Percentage Change in Spectral-domain Optical Coherence Tomography (SD-OCT) Average Retinal Nerve Fiber Layer (RNFL) Thickness at baseline and every year. | baseline, year1, year2, year3, year4, year5.
  Adjusted mean percentage change in thickness of the RNFL every year for the affected eye from the baseline as determined by SD-OCT.
Percentage change in SD-OCT Average Retinal Ganglion Cell Layer/Inner Plexiform Retinal Layer (RGCL/IPL) every year. | baseline, year1, year2, year3, year4, year5.
  Adjusted mean change in thicknesses of the RGCL/IPL every year for the affected eye from the baseline as determined by segmentation of SD-OCT.
Changes in cognitive function of patients with IDD at baseline and over time during follow-up | baseline, year1, year2, year3, year4, year5.
  Scale assessment mainly rely on SDMT(Symbol Digit Modalities Test), MoCA( Montreal Cognitive Assessment), MMSE(Mini-mental State Examination) and so on. The Symbol Digit Modalities Test (SDMT) is widely used because it is easy to administer, reliable and also evaluates information processing speed. The Montreal Cognitive Assessment (MoCA) is a brief, 30-question test that helps healthcare professionals detect cognitive impairments very early on, allowing for faster diagnosis and patient care. The Mini-Mental State Exam (MMSE) is a widely used test of cognitive function among the elderly; it includes tests of orientation, attention, memory, language and visual-spatial skills.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | From baseline to 5 years
  Treatment-emergent adverse events, treatment-emergent serious adverse events (TESAEs), including laboratory measurements as well as their changes or shift from baseline over time
NF-L level in serum. | baseline, year1, year2, year3, year4, year5.
  Neurofilament light (NF-L) is a 68 kDa cytoskeletal intermediate filament protein that is expressed in neurons. Elevated blood concentrations of neurofilament light chain (NfL) were found to correlate with an increase in the number of relapses, disability worsening, MRI disease activity, and brain volume loss in MS.
Determination of serum autoimmune antibodies | baseline, year1, year2, year3, year4, year5.
  Compare serum AQP4(Aquaporin 4)-ab titers, MOG(Myelin Oligodendrocyte Glycoprotein)-ab titers, MBP(myelin basic protein)-ab titers at baseline and every year.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Xu Y, Meng H, Fan M, Yin L, Sun J, Yao Y, Wei Y, Cong H, Wang H, Song T, Yang CS, Feng J, Shi FD, Zhang X, Tian DC. A Simple Score (MOG-AR) to Identify Individuals at High Risk of Relapse After MOGAD Attack. Neurol Neuroimmunol Neuroinflamm. 2024 Nov;11(6):e200309. doi: 10.1212/NXI.0000000000200309. Epub 2024 Sep 9. PMID 39250723